CLINICAL TRIAL: NCT00070616
Title: An Open-label Study of the Pharmacokinetics (PK) of Recombinant Human Keratinocyte Growth Factor (Palifermin; rHuKGF) in Subjects With Hematologic Malignancies Undergoing Total Body Irradiation and High-dose Chemotherapy Followed by Peripheral Blood Progenitor Cell (PBPC) Transplantation
Brief Title: Pharmacokinetic Study of Palifermin in Subjects Receiving Radiation Therapy and Chemotherapy Followed by Blood Stem Cell Support
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20010182; NCT00963170 (obsolete NCT alias)
Record Dates: First submitted 2003-10-06; First posted 2003-10-08 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Leukemia; Lymphoma; Myeloma
Keywords: mucositis; chemotherapy; radiation therapy
MeSH Terms: conditions — Leukemia; Lymphoma; Neoplasms, Plasma Cell; Mucositis | interventions — Radiotherapy; Drug Therapy

ARMS (2):
- Palifermin 6 x 60 μg/kg/day (Experimental): The first 3 consecutive daily doses were administered before the initiation of conditioning therapy (study days -11, -10, and -9); 3 additional consecutive daily doses were administered after administration of radiotherapy, chemotherapy and PBPC transplantation (study days 0, 1, and 2).
  Interventions: Drug: Palifermin 6 x 60 μg/kg/day; Radiation: radiotherapy; Drug: Chemotherapy
- Palifermin 2 x 180 μg/kg/day (Experimental): The first dose was administered on study day -11, 3 days before the initiation of conditioning therapy, and the second dose was given on day 0 after administration of radiotherapy, chemotherapy and the PBPC infusion
  Interventions: Drug: Palifermin 2 x 180 μg/kg/day; Radiation: radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Drug: Palifermin 6 x 60 μg/kg/day
  Arms: Palifermin 6 x 60 μg/kg/day
Drug: Palifermin 2 x 180 μg/kg/day
  Arms: Palifermin 2 x 180 μg/kg/day
Radiation: radiotherapy
Drug: Chemotherapy

SUMMARY:
Open label palifermin will be administered to subjects who are at a risk of developing mucositis after radiotherapy and chemotherapy followed by blood stem cell support. The amount of palifermin in the blood following administration will be evaluated. The safety of palifermin administration and its effect on reducing mucositis will also be evaluated.

DETAILED DESCRIPTION:
Mucositis is a common side effect to chemotherapy and radiotherapy involving the formation of erythema and ulcerative lesions in the mouth. Mucositis can be serious, resulting in pain requiring interventions such as analgesic medications and the use of parenteral feedings. Currently, no standard therapy is available to prevent or treat mucositis.

ELIGIBILITY:
* Patients diagnosed with Non-Hodgkin's Lymphoma, Hodgkin's Disease, Leukemia and Myeloma. - Eligible for treatment with radiation therapy and chemotherapy followed by blood stem cell support.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
To characterize the PK profile of 3 daily intravenous (IV) doses of rHuKGF before total body irradiation (TBI) / high-dose chemotherapy conditioning treatment and after PBPC transplantation

SECONDARY OUTCOMES:
To assess the safety and tolerability of rHuKGF in subjects with hematologic malignancies undergoing TBI and high-dose chemotherapy followed by PBPC transplantation.
To assess oral mucositis in subjects receiving rHuKGF.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Zia-Amirhosseini P, Hurd DD, Salfi M, Cheah TC, Aycock J, Cesano A. Pharmacokinetics of palifermin administered as the standard dose and as a collapsed dose in patients with hematologic malignancies. Pharmacotherapy. 2007 Oct;27(10):1353-60. doi: 10.1592/phco.27.10.1353. PMID 17896890
- See also: FDA-approved Drug Labeling — http://www.kepivance.com/